CLINICAL TRIAL: NCT03148379
Title: A Multi-center, Prospective, Randomized Study Comparing Surgical and Economic Parameters of Total Knee Replacement Performed With Single-use Efficiency Instruments With Patient Specific Technique (MyKnee®) Versus Traditional Metal Instruments With Conventional Surgical Technique.
Brief Title: Single-use Efficiency Instruments With Patient Specific Technique (MyKnee®) Versus Traditional Metal Instruments With Conventional Surgical Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20161119
Record Dates: First submitted 2017-04-20; First posted 2017-05-11 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis
Keywords: Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Customized patient instruments (Experimental): Experimental group: Patients randomized into this group will undergo surgery utilizing single-use Efficiency Instruments with patient-specific technique (MyKnee® patient-matched cutting blocks)
  Interventions: Device: Customized patient instruments
- Traditional metal instruments (Active Comparator): Control Group: Patients will undergo conventional surgical technique
  Interventions: Device: Traditional Metal Instruments

INTERVENTIONS:
Device: Customized patient instruments — Single use efficiency instruments and cutting blocks specifically made for each patient using pre-op MRI or CT scans to make bone cuts and select implant size.
  Other Names: Single-use Efficiency Instruments with Patient Specific Technique (MyKnee®)
  Arms: Customized patient instruments
Device: Traditional Metal Instruments — Traditional metal instrument will be used to make bone cuts and size the components in this control group.
  Other Names: Traditional Metal Instruments with Conventional Surgical Technique
  Arms: Traditional metal instruments

SUMMARY:
To compare economic factors and the rate of adverse events between two types of instrumentation used for total knee replacement: Single-use Efficiency Instruments with Patient Specific Technique (MyKnee®) Traditional Metal Instruments with Conventional Surgical Technique

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* BMI ≤35
* Undergoing unilateral total knee arthroplasty due to osteoarthritis (primary or post-traumatic OA)
* Able and willing to give consent and to comply with study requirements, including follow up visit at 6 weeks

Exclusion Criteria:

* Pregnant women or those seeking to become pregnant. Pregnancy test is administered prior to surgery as part of routine care by the hospital / surgery center for all female patients of childbearing potential
* Is participating in another clinical study
* Has inflammatory arthritis
* Has knee avascular necrosis
* Has severe deformity, defined as greater than 10 degrees varus or valgus relative to the mechanical axis
* Has retained hardware in the knee that requires removal or interferes with Total Knee Arthroplasty (TKA) procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh Ahuja, MBBS, MS, Study Director — Medacta USA
Locations (5):
- United States (5):
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Ortho Montana, Billings, Montana
  - Orthopedic Associates Meadville, Meadville, Pennsylvania
  - Texas Orthopedics, Austin, Texas
  - Jordan Valley Medical Center of Orthopedics Rehabilitation and Excellence, West Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Started | 21 | 11
Completed | 20 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments | Total
Number analyzed (Participants) | 21 | 11 | 32
Age, Continuous [Mean (Full Range); unit: years] | 67.24 [56 to 75] | 65 [53 to 70] | 66.47 [53 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 15 | 3 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 21 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: OR Total Time
Description: Total time patient is in operating room
Time Frame: Day of Surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
minutes | 93.00 [81.90 to 113.27] | 92.72 [82.73 to 101.00]

2. Primary Outcome: Opening Instruments
Description: Time to open surgical instruments
Time Frame: Day of Surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
minutes | 8.23 [4.20 to 33.50] | 7.42 [3.70 to 14.00]

3. Primary Outcome: Back Table Setup Time
Description: Time to set up back surgical table
Time Frame: Day of Surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
minutes | 21.33 [5.68 to 31.32] | 21.62 [1.42 to 37.73]

4. Primary Outcome: Tourniquet Time
Description: Time tourniquet is on patient during surgery
Time Frame: Day of Surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
minutes | 58.75 [47.43 to 76.48] | 58.25 [46.07 to 72.13]

5. Primary Outcome: Incision to Skin Closure
Description: Time from incision to skin closure during surgery
Time Frame: Day of Surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
minutes | 55.37 [41.77 to 112.92] | 55.03 [43.57 to 63.87]

6. Primary Outcome: Bone Prep Time
Description: Time to prepare bone for implant during surgery
Time Frame: Day of Surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
minutes | 17.83 [12.47 to 32.78] | 17.67 [9.95 to 17.87]

7. Primary Outcome: Patella Resection Time
Description: Time to resection patella during surgery
Time Frame: Day of Surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
minutes | 2.27 [0.83 to 5.93] | 2.22 [1.18 to 3.32]

8. Primary Outcome: Clean-up Time
Description: Time to clean up following surgery
Time Frame: Day of Surgery
Measure: Mean (Full Range); unit: minutes
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
minutes | 7.67 [1.48 to 20.98] | 8.40 [1.37 to 24.13]

9. Secondary Outcome: Hemoglobin Range
Description: Post op 1 day hemoglobin range
Time Frame: 24 hours or at discharge if patient does not stay overnight
Measure: Mean (Full Range); unit: grams per deciliter (g/dl)
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
grams per deciliter (g/dl) | 13.3 [8.9 to 18.1] | 13.3 [11.5 to 15.8]

10. Secondary Outcome: Surgical Waste Weight
Description: Weigh surgical waste at the end of each surgery
Time Frame: Day of Surgery
Measure: Mean (Full Range); unit: pounds
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
pounds | 29.8 [21.0 to 35.3] | 21.1 [17.6 to 23.9]

11. Secondary Outcome: Mechanical Axis
Description: Radiographic analysis of mechanical axis alignment
Time Frame: Pre-Operative
Measure: Mean (Full Range); unit: degrees
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
degrees | 175.5 [165.9 to 186.6] | 175.85 [168.1 to 184.4]

12. Secondary Outcome: Mechanical Axis
Description: Radiographic analysis of mechanical axis alignment
Time Frame: Post-Operative
Measure: Mean (Full Range); unit: degrees
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 20 | 11
degrees | 78.4 [0.0 to 179.5] | 72.6 [0.8 to 186.0]

13. Secondary Outcome: Tibial Slope
Description: Radiographic analysis of Tibial Posterior Slope
Time Frame: Pre-Operative
Measure: Mean (Full Range); unit: degrees
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 21 | 11
degrees | 7.6 [2.0 to 12.0] | 7.6 [3.0 to 12.0]

14. Secondary Outcome: Tibial Slope
Description: Radiographic analysis of Tibial Posterior Slope
Time Frame: Post-Operative
Measure: Mean (Full Range); unit: degrees
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
Number analyzed (Participants) | 20 | 11
degrees | 4.3 [0.0 to 6.5] | 4.2 [2.7 to 8.4]

ADVERSE EVENTS:
Time Frame: Surgery to 6 weeks post-op
Arm/Group | Customized Patient Instruments | Traditional Metal Instruments
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/11
Other Adverse Events (participants affected / at risk) | 0/21 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT03148379/Prot_SAP_000.pdf